CLINICAL TRIAL: NCT00884546
Title: A Phase Ib Multiple Ascending Dose Study of BMS-833923 Alone or in Combination With Lenalidomide (Revlimid) Plus Dexamethasone or in Combination With Bortezomib (Velcade) in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Multiple Ascending Dose (MAD) Combination in Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA194-003
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancer, Various, NOS
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic | interventions — BMS-833923; Lenalidomide; Dexamethasone; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): BMS-833923 (Starting dose is a loading dose of 60 mg for 7 days with a 30 mg daily dose thereafter)
  Interventions: Drug: BMS-833923
- Arm 2 (Active Comparator): BMS-833923 (MTD or below)
  Lenalidomide (at or below the recommended prescribing dose)
  Dexamethasone (40 mg)
  Interventions: Drug: BMS-833923; Drug: Lenalidomide; Drug: Dexamethasone
- Arm 3 (Active Comparator): BMS-833923 (MTD or below)
  Bortezomib (at or below the recommended prescribing dose)
  Interventions: Drug: BMS-833923; Drug: Bortezomib

INTERVENTIONS:
Drug: BMS-833923 — Capsule, Oral, Once daily, 6 months
Drug: Lenalidomide — Capsule, Oral, Once daily, 6 months
  Other Names: Revlimid
  Arms: Arm 2
Drug: Dexamethasone — Capsule, Oral, Once a week, 6 months
  Arms: Arm 2
Drug: Bortezomib — Powder, IV, On days 1, 4, 8, 11, 6 months
  Other Names: Velcade
  Arms: Arm 3

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of BMS-833923 administered alone, in combination with lenalidomide plus dexamethasone, or in combination with bortezomib in subjects with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Multiple Myeloma
* Men and Women at least 18 years old
* ECOG status 0-2
* Last therapeutic or diagnostic treatment at least 21 days prior
* Bone marrow transplants must have been completed at least 3 months prior
* Any toxicity from prior therapies must have resolved to Grade ≤1

Exclusion Criteria:

* Women pregnant or breastfeeding
* WOCBP unwilling/unable to use acceptable method to avoid pregnancy
* Uncontrolled medical disorder or active infection
* Current or recent (w/in 3 months) gastrointestinal disorder
* Inability to swallow oral medication
* Inability to be venipunctured
* Uncontrolled or significant cardiovascular disease
* Uncontrolled hyperlipidemia
* Intolerance of lenalidomide or bortezomib if participating in Arms B and C
* Concurrent therapy with any other investigational product
* Subjects involuntary incarcerated
* Subjects detained for treatment of psychiatric or physical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To establish DLT(s), MTD, and Phase 2 dose range and schedule of BMS-833923 administered alone, in combination with two dose levels of lenalidomide plus dexamethasone, or with two dose levels of bortezomib in subjects with relapsed or refractory MM | For Treatment Arms A and B, outcome would be measured for approximately 5 months on Days 1, 8, 15, and 28 for Cycles 1 and 2 and then every 28 days for the following cycles

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of BMS-833923 as a single agent or in combination with two dose levels of lenalidomide plus a fixed low-dose of dexamethasone or in combination with two dose levels of bortezomib | For Treatment Arms A and B, outcome would be measured for approximately 5 months on Days 1, 8, 15, and 28 for Cycles 1 and 2 and then every 28 days for the following cycles
To evaluate the Pharmacokinetics of BMS-833923 | For Treatment Arms A and B, outcome would be measured for approximately 5 months on Days 1, 8, 15, and 28 for Cycles 1 and 2 and then every 28 days for the following cycles
To evaluate the Pharmacodynamics effects of BMS-833923 | For Treatment Arms A and B, outcome would be measured for approximately 5 months on Days 1, 8, 15, and 28 for Cycles 1 and 2 and then every 28 days for the following cycles

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (8):
  - City Of Hope National Medical Center, Duarte, California
  - Moores Ucsd Cancer Center, La Jolla, California
  - Local Institution, Los Angeles, California
  - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Local Institution, Detroit, Michigan
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Oncology Consultants, Pa, Houston, Texas
  - Cancer Therapy And Research Center, San Antonio, Texas

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx